CLINICAL TRIAL: NCT02734810
Title: A Phase 3, Open-Label Study Evaluating the Efficacy and Safety of Liprotamase in Subjects With Cystic Fibrosis-Related Exocrine Pancreatic Insufficiency
Brief Title: SIMPLICITY: Studying Impacts on Malabsorption With Liprotamase in Cystic Fibrosis
Acronym: SIMPLICITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN-EPI3332
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
Keywords: Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Liprotamase; Pancreatic Enzyme Replacement Therapy (PERT)
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — Solutions; liprotamase lipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Liprotamase Powder for Oral Solution in Subjects aged ≥7 years of age
  Interventions: Drug: Liprotamase Powder for Oral Solution
- Part B (Experimental): Liprotamase Powder for Oral Solution in Subjects aged 28 days to <7 years
  Interventions: Drug: Liprotamase Powder for Oral Solution

INTERVENTIONS:
Drug: Liprotamase Powder for Oral Solution — Oral, soluble, non-enterically coated, non-porcine, pancreatic enzyme replacement therapy
  Other Names: Liprotamase

SUMMARY:
Liprotamase consists of 3 soluble, non-porcine digestive enzymes, lipase, protease, and amylase, combined in a fixed ratio. Liprotamase is stable in the stomach and can be formulated without enteric coating for administration either as a capsule or as a dosing solution dissolved in water or juice. The purpose of the present study is to provide efficacy and safety data for a new, soluble formulation of liprotamase, Liprotamase Powder for Oral Solution, in Cystic Fibrosis patients with exocrine pancreatic insufficiency (EPI).

ELIGIBILITY:
Inclusion Criteria:

* For Part A: males or females ≥7 years of age
* For Part B: males or females 28 days to <7 years
* Diagnosis of cystic fibrosis based on presentation, genotype and/or sweat chloride
* Low fecal elastase
* Fair-to-good nutritional status

Exclusion Criteria:

* History or diagnosis of fibrosing colonopathy
* Distal intestinal obstruction syndrome in 6 months prior to screening
* Receiving enteral tube feedings
* Chronic diarrheal illness unrelated to pancreatic insufficiency
* Liver abnormalities, or liver or lung transplant, or significant bowel resection

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Investigator Site 139, Little Rock, Arkansas
  - Investigator Site, Orange, California
  - Investigator Site 114, Aurora, Colorado
  - Investigator Site 117, Altamonte Springs, Florida
  - Investigator Site 138, Hollywood, Florida
  - Investigator Site 130, Miami, Florida
  - Investigator Site 110, Atlanta, Georgia
  - Investigator Site 109, Glenview, Illinois
  - Investigator Site 105, Wichita, Kansas
  - Investigator Site 122, Louisville, Kentucky
  - Investigator Site 132, Portland, Maine
  - Investigator Site 124, Ann Arbor, Michigan
  - Investigator Site 135, Las Vegas, Nevada
  - Investigator Site 118, Durham, North Carolina
  - Investigator Site 101, Oklahoma City, Oklahoma
  - Investigator Site 136, Oklahoma City, Oklahoma
  - Investigator Site 106, Hershey, Pennsylvania
  - Investigator Site 111, Dallas, Texas
  - Investigator Site 116, Houston, Texas
  - Investigator Site 112, Richmond, Virginia
  - Investigator Site 129, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A | Part B
Started | 15 | 0
Completed | 13 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 15 | 0 | 15
Age, Continuous [Mean (Full Range); unit: years] | 24.1 [8 to 52] |  | 24.1 [8 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 12 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 0 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Number of subjects reporting 1 or more adverse events
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 15 | 0
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/0
Other Adverse Events (participants affected / at risk) | 3/15 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=15) | Part B (N=0)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=15) | Part B (N=0)
Infective exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other